CLINICAL TRIAL: NCT00881621
Title: Phase II Study of Lapatinib and Capecitabine in 2nd Line Treatment of Locally Advanced/Metastatic Pancreatic Cancer
Brief Title: Lapatinib and Capecitabine for Second Line Treatment of Pancreas Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Georgetown University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 011438; IND #103,981 (Other: FDA); 2008-437 (Other: IRB)
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2017-01

CONDITIONS: Pancreas Cancer
Keywords: Pancreas cancer; lapatinib; capecitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib and Capecitabine (Experimental): Treatment
  Interventions: Drug: Lapatinib and Capecitabine

INTERVENTIONS:
Drug: Lapatinib and Capecitabine — Lapatinib 1250-mg PO daily one hour before or after meals Capecitabine 1000 mg/m2 PO twice daily on days 1-14 of 21-day cycle for a total of 8 cycles
  Other Names: Tykerb; GW572016

SUMMARY:
Patients are being asked to participate in this study who have locally advanced or metastatic pancreatic cancer (cancer of the pancreas that has spread to another part of the body) that has gotten worse after first-line chemotherapy.

The purpose of this study is to see if the drugs, Capecitabine and Lapatinib (two chemotherapy agents), prolong survival and improve quality of life as compared to supportive care alone.

Lapatinib in combination with a drug called capecitabine, has been approved by the Food and Drug Administration (FDA) for the treatment of metastatic breast cancer. It has not yet been approved to treat this type of cancer. Both of these drugs are pills.

This research is being done because it is not known if the combination of Capecitabine and Lapatinib is better than supportive care alone for pancreatic cancer.

DETAILED DESCRIPTION:
This is an open-label single-arm Phase II trial for patients with metastatic pancreatic cancer who have failed first line Gemcitabine-based therapy. Patients will be treated with a combination of Capecitabine and Lapatinib, a dual tyrosine-kinase inhibitor of EGFR and HER-2.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the pancreas
* Prior failed 1st line gemcitabine therapy for metastatic disease or relapsed within six months of completion of gemcitabine adjuvant therapy
* Prior capecitabine or 5fu is allowed in the setting of radiation
* Must either be able to swallow or receive enteral nutrition via gastrostomy feeding tube
* Cardiac ejection fraction within institutional range of normal as measured by echocardiogram
* ECOG performance status 0-2
* Signed informed consent form
* Adequate hepatic, bone marrow, and renal function

Exclusion Criteria:

* Any prior treatment with lapatinib, or any anti-HER2 treatment or any anti-EGFR treatment
* Not recovered from adverse events to a toxicity grade </= 1 due to prior chemotherapy
* More than one prior chemotherapy regimens
* Known brain metastases, uncontrolled seizure disorders, encephalitis, or multiple sclerosis
* HIV positive on antiretroviral therapy
* Pregnant or lactating
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib or capecitabine
* Malabsorption syndrome or uncontrolled inflammatory GI disease (Crohn's or ulcerative colitis)
* Known history of uncontrolled or symptomatic angina, arrhythmia, or congestive heart failure
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/ social situations that would limit compliance with study requirements
* Known dihydropyrimidine dehydrogenase deficiency
* Concurrent malignancy unless the subject has been curatively treated and disease free for >/= 2 years or the cancer was non-melanoma skin cancer or early cervical cancer.
* Creatinine clearance < 30 mL/min
* Absolute neutrophil count < 1500, platelets < 75,000
* Transaminases > 3.0 times the upper limit of normal, except in known hepatic metastasis, wherein they must be < 5.0 times the upper limit of normal
* Total bilirubin > 1.5 times the ULN, > 2.5 x ULN if patient has Gilbert's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-08; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth He, MD, PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to change of practice, it is difficult to complete the enrollment for the study
Period: Overall Study
Arm/Group | Lapatinib and Capecitabine
Started | 51
Completed | 17
Not Completed | 34
Not completed — Physician Decision | 34

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib and Capecitabine
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
ECOG [Number; unit: participants] — ECOG PERFORMANCE STATUS* Grade 0: Fully active, able to carry on all pre-disease performance without restriction
  1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work 2: Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours 4: Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair 5: Dead
  participants
    ECOG PS 0 | 3
    ECOG PS 1 | 12
    ECOG PS2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time of study entry to time of death
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib and Capecitabine
Number analyzed (Participants) | 17
months | 5.2 [3.4 to 9]

2. Secondary Outcome: Clinical Benefit Response
Description: number of participants who had stable disease or partial response or complete response per Response Evaluation Criteria In Solid Tumors.
  Complete Response: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Stable Disease: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Lapatinib and Capecitabine
Number analyzed (Participants) | 17
participants | 6

3. Secondary Outcome: Progression Free Survival
Description: Time of study entry to cancer progression.
Time Frame: 24 months
Population: Time of study entry to disease progression.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib and Capecitabine
Number analyzed (Participants) | 17
months | 2.6 [1.3 to 3.8]

4. Secondary Outcome: Adverse Events
Description: Grade 3 or 4 toxicities
Time Frame: 2 years
Population: grade 3 or 4 toxicities
Measure: Number; unit: participants
Arm/Group | Lapatinib and Capecitabine
Number analyzed (Participants) | 17
participants | 3

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Lapatinib and Capecitabine
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib and Capecitabine (N=17)
fatigue (General disorders) | 1 (1)
nausea, vomiting (Gastrointestinal disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib and Capecitabine (N=17)
fatigue (General disorders) | 7 (7)
anorexia (General disorders) | 1 (1)
nausea vomiting (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 5 (5)
hand-foot syndrome (Skin and subcutaneous tissue disorders) | 3 (3)
skin rash (Skin and subcutaneous tissue disorders) | 2 (2)
sensort neuropathy (Nervous system disorders) | 1 (1)
stomatitis (Gastrointestinal disorders) | 2 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less